CLINICAL TRIAL: NCT02255461
Title: Phase I Study of CDK 4-6 Inhibitor PD-0332991 (Palbociclib; IBRANCE) in Children With Recurrent, Progressive or Refractory Central Nervous System Tumors
Brief Title: Palbociclib Isethionate in Treating Younger Patients With Recurrent, Progressive, or Refractory Central Nervous System Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Data for the primary objectives is complete and the MTD identified in Stratum II.
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBTC-042; U01CA081457 (NIH)
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Results first posted 2020-04-08 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Childhood Choroid Plexus Tumor; Childhood Ependymoblastoma; Childhood Grade III Meningioma; Childhood High-grade Cerebellar Astrocytoma; Childhood High-grade Cerebral Astrocytoma; Childhood Medulloepithelioma; Recurrent Childhood Anaplastic Astrocytoma; Recurrent Childhood Anaplastic Oligoastrocytoma; Recurrent Childhood Anaplastic Oligodendroglioma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Cerebellar Astrocytoma; Recurrent Childhood Cerebral Astrocytoma; Recurrent Childhood Giant Cell Glioblastoma; Recurrent Childhood Glioblastoma; Recurrent Childhood Gliomatosis Cerebri; Recurrent Childhood Gliosarcoma; Recurrent Childhood Medulloblastoma; Recurrent Childhood Pineoblastoma; Recurrent Childhood Supratentorial Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Choroid Plexus Neoplasms; Astrocytoma; Oligodendroglioma; Glioblastoma; Neoplasms, Neuroepithelial; Medulloblastoma | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Treatment (palbociclib isethionate) (Experimental): Patients receive palbociclib isethionate PO QD on days 1-21. Treatment repeats every 4 weeks for 26 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: palbociclib isethionate; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: palbociclib isethionate — Given PO
  Other Names: 6-acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)pyrido[2,3-d]pyrimidin-7(8H)-one, 827022-33-3, palbociclib, PD 0332991-0054, PD-0332991, PD-332991, PF-00080665-73
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of palbociclib isethionate in treating younger patients with central nervous system tumors that have grown, come back, or not responded to treatment. Palbociclib isethionate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD)/phase II recommended dose and describe toxicities related to PD-0332991 (palbociclib isethionate) in children with retinoblastoma protein 1 (Rb1) positive recurrent, progressive or refractory primary central nervous system (CNS) tumors.

II. To determine plasma pharmacokinetics of PD-0332991 in children with Rb1positive recurrent, progressive or refractory primary CNS tumors.

SECONDARY OBJECTIVES:

I. To record preliminary evidence of efficacy of PD-0332991 in children with recurrent CNS tumors.

II. To evaluate cyclin-dependent kinase (CDK)4/6, cyclin D1-3, Ink4a-ARF copy-number variations in available tumor tissue by array comparative, genomic hybridization (aCGH).

III. To explore the potential relationships between the pharmacokinetics of PD-0332991 and pharmacodynamic response (e.g. percentage change in absolute neutrophil count [ANC], platelet counts).

IV. To explore the pharmacogenetic polymorphisms in PD-0332991 metabolizing enzymes and transporters and relate these polymorphisms to PD-0332991 pharmacokinetics.

OUTLINE: This is a dose-escalation study.

Patients receive palbociclib isethionate orally (PO) once daily (QD) on days 1-21. Treatment repeats every 4 weeks for 26 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with retinoblastoma protein (Rb1) positive recurrent, progressive or refractory central nervous system (CNS) tumors
* Histologically confirmed Rb1 positive primary recurrent, progressive, or refractory central nervous system tumors; patients with low grade gliomas are excluded
* Formalin fixed paraffin embedded tumor tissue (preferably from current recurrence) must be available to assess Rb1 protein status prior to enrollment; only patients with recurrent diffuse intrinsic brain stem glioma (DIPG) can be enrolled without the need for available tumor tissue for Rb1 protein status confirmation
* Patients must have measurable disease (in 2-dimensions) on magnetic resonance imaging (MRI) scan of brain and/or spine to assess preliminary evidence of response
* Body surface area (BSA):

  * Patients enrolled on dose level 1 (50 mg/m^2) must have BSA >= 1.20 m^2
  * Patients enrolled on dose level 2 (75 mg/m^2) must have BSA >= 0.93 m^2
  * Patients enrolled on dose level 3 (95 mg/m^2) must have BSA >= 0.70 m^2
* Patients must have received no more than 2 prior chemotherapy regimens and/or focal radiotherapy for their brain tumor and fully recovered from the acute treatment related toxicities of all prior therapies prior to entering this study; for those acute baseline adverse events attributable to prior therapy, patients must meet organ function criteria
* Chemotherapy: patients must have received their last dose of known myelosuppressive anticancer chemotherapy at least three (3) weeks prior to study enrollment in the study or at least six (6) weeks for those receiving nitrosourea
* Biologic therapy: patients should have received their last dose of biologic agent >= 7 days prior to enrollment; in the event the patient has received another biologic agent and has experienced >= grade 2 myelosuppression, then at least three (3) weeks must have elapsed prior to enrollment; if the investigational or biologic agent has a prolonged half-life then at least three (3) weeks interval is required
* Radiotherapy: patients must have had their last fraction of:

  * Focal irradiation > 2 weeks prior to enrollment
* Corticosteroids: patients who are receiving dexamethasone or other corticosteroids must be on a stable or decreasing dose for at least 1 week prior to enrollment; it is recommended that patients be off all steroid therapy or receive the least dose that will control their neurologic symptoms
* Growth factors: all colony forming growth factor(s) have been discontinued for at least one week prior to enrollment (filgrastim, sargramostim, and erythropoietin); for patients on long acting growth factors, the interval should be two weeks
* Patients with neurological deficits that are stable for a minimum of one week prior to registration
* Patients must be able to swallow capsules
* Karnofsky performance scale (KPS for > 16 years of age) or Lansky performance score (LPS for =< 16 years of age) assessed within two weeks of enrollment must be >= 60
* Absolute neutrophil count >= 1,000/mm^3
* Platelets >= 100,000/mm^3 transfusion independent (no platelet transfusion one week prior to enrollment)
* Hemoglobin >= 8 g/dl
* Total bilirubin =< 1.5 times upper limit of institutional normal (ULN) for age
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal for age
* Serum albumin >= 3 g/dL
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * 1 to < 2 years: 0.6 (male), 0.6 (female)
  * 2 to < 6 years: 0.8 (male), 0.8 (female)
  * 6 to < 10 years: 1 (male), 1 (female)
  * 10 to < 13 years: 1.2 (male), 1.2 (female)
  * 13 to < 16 years: 1.5 (male), 1.4 (female)
  * >= 16 years: 1.7 (male), 1.4 (female)
* Female patients of childbearing potential must have a negative serum pregnancy test at the time of enrollment
* Patients of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control while being treated on this study
* Patient and/or guardian have the ability to understand and the willingness to sign a written informed consent document according to institutional guidelines

Exclusion Criteria:

* Patients with any clinical significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction) that is likely to interfere with the study procedures or results
* Patients with low grade gliomas and Rb1 negative tumors
* Patients who have received any of the following:

  * > 2 chemotherapy regimens
  * Myeloablative chemotherapy with stem cell rescue
  * Craniospinal irradiation
* Patients with corrected QT (QTc) interval of > 450 msec or those on medications known to prolong QTc interval
* Prior treatment on a CDK inhibitor
* Patients who are receiving drugs that are strong inducers or inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4)
* Patients who are receiving any other investigational therapy
* Patients who require enzyme inducing anti-convulsants to control seizures
* Patients with cataracts on ophthalmologic examination

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Van Mater, MD, Principal Investigator — Pediatric Brain Tumor Consortium
Locations (11):
- United States (11):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children Hospital Stanford University, Palo Alto, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Lurie Childrens Hospital-Chicago, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children Hospital Medical Center, Cincinnati, Ohio
  - Children Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children Research Hospital, Memphis, Tennessee
  - Texas Childrens Hospital, Houston, Texas
  - Seattle Children Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raetz EA, Teachey DT, Minard C, Liu X, Norris RE, Denic KZ, Reid J, Evensen NA, Gore L, Fox E, Loh ML, Weigel BJ, Carroll WL. Palbociclib in combination with chemotherapy in pediatric and young adult patients with relapsed/refractory acute lymphoblastic leukemia and lymphoma: A Children's Oncology Group study (AINV18P1). Pediatr Blood Cancer. 2023 Nov;70(11):e30609. doi: 10.1002/pbc.30609. Epub 2023 Aug 8. PMID 37553297

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients between 4 and 21 years of age with histologically confirmed retinoblastoma protein (Rb1) positive, primary recurrent, progressive, or refractory central nervous system tumors were enrolled at Pediatric Brain Tumor Consortium member institutions. The first patient was enrolled on 12/8/2014 and the last patient was enrolled on 10/10/2018.
Pre-assignment Details: All 35 eligible patients enrolled were included. The 'Completed' row included patients who completed all protocol therapy or who experienced a protocol endpoint which took them off therapy. These included dose limiting toxicities and progression/relapse events. Adverse events not related to study agent were included in the 'Not Completed' row.
Groups:
- Stratum I, Dose Level 1 (50 mg/m2): Less-heavily pre-treated patients received oral palbociclib daily at 50 mg/m2/day for 21 days followed by a week rest (one course = 28 days) for up to 26 courses in the absence of disease progression or unacceptable toxicity.
- Stratum I, Dose Level 2 (75 mg/m2): Less-heavily pre-treated patients received oral palbociclib daily at 75 mg/m2/day for 21 days followed by a week rest (one course = 28 days) for up to 26 courses in the absence of disease progression or unacceptable toxicity.
- Stratum I, Dose Level 3 (95 mg/m2): Less-heavily pre-treated patients received oral palbociclib daily at 95 mg/m2/day for 21 days followed by a week rest (one course = 28 days) for up to 26 courses in the absence of disease progression or unacceptable toxicity.
- Stratum II, Dose Level 1 (50 mg/m2): Heavily pre-treated patients received oral palbociclib daily at 50 mg/m2/day for 21 days followed by a week rest (one course = 28 days) for up to 26 courses in the absence of disease progression or unacceptable toxicity.
- Stratum II, Dose Level 2 (75mg/m2): Heavily pre-treated patients received oral palbociclib daily at 75 mg/m2/day for 21 days followed by a week rest (one course = 28 days) for up to 26 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2)
Started | 3 | 12 | 6 | 4 | 10
Completed | 3 | 10 | 5 | 4 | 8
Not Completed | 0 | 2 | 1 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1
Not completed — Not meet dose reduction BSA requirement | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Summary statistics for baseline characteristics are shown for all enrolled patients (n = 35).
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2) | Total
Number analyzed (Participants) | 3 | 12 | 6 | 4 | 10 | 35
Age, Continuous [Median (Full Range); unit: years] | 16.6 [9.7 to 16.6] | 12.6 [7.0 to 21.1] | 9.3 [4.9 to 19.3] | 16.5 [13.3 to 17.2] | 10.5 [6.3 to 21.6] | 12.7 [4.9 to 21.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 3 | 0 | 3 | 12
  Male | 2 | 7 | 3 | 4 | 7 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 2 | 0 | 3 | 8
  Not Hispanic or Latino | 3 | 6 | 4 | 2 | 5 | 20
  Unknown or Not Reported | 0 | 3 | 0 | 2 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 1 | 1 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 2 | 4
  White | 2 | 7 | 4 | 3 | 7 | 23
  More than one race | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 12 | 6 | 4 | 10 | 35

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Palbociclib in Stratum I
Description: Rolling-6 design was used to estimate MTD. The MTD was empirically defined as the highest dose level at which six patients were treated with at most one patient experiencing a dose-limiting toxicity (DLT) and the next higher dose level had been determined to be too toxic. Stratum I consisted of less-heavily pre-treated patients.
Time Frame: 4 weeks
Population: Patients who were enrolled on stratum I and were evaluable for dose finding assessment were used to determine the MTD for stratum I.
Measure: Number; unit: mg/m2/day
Groups:
- Stratum I: Of 21 patients enrolled on stratum I, 2 patients were not evaluable for dose finding assessment due to receiving less than required dose of study drug. The remaining 19 patients were used to determine the MTD for stratum I.
Arm/Group | Stratum I
Number analyzed (Participants) | 19
mg/m2/day | 75

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Palbociclib in Stratum II
Description: Rolling-6 design was used to estimate MTD. The MTD was empirically defined as the highest dose level at which six patients were treated with at most one patient experiencing a DLT and the next higher dose level had been determined to be too toxic. Stratum II consisted of heavily pre-treated patients.
Time Frame: 4 weeks
Population: Patients who were enrolled on stratum II and were evaluable for dose finding assessment were used to determine the MTD for stratum II.
Measure: Number; unit: mg/m2/day
Groups:
- Stratum II: Of 14 patients enrolled on stratum II, 3 patients were not evaluable for dose finding assessment: 2 patients due to receiving less than required dose of study drug and 1 due to withdrawal consent prior to beginning protocol therapy. The remaining 11 patients were used to determine the MTD for stratum II.
Arm/Group | Stratum II
Number analyzed (Participants) | 11
mg/m2/day | 75

3. Primary Outcome: Number of Patients Who Experienced Dose Limiting Toxicities (DLTs)
Description: DLTs were defined as any of the following adverse events that were at least possibly related to palbociclib that occurred during the first 4 weeks of therapy regardless of expectedness. Hematologic DLTs included grade 3 neutropenia with fever and sepsis, grade 3 thrombocytopenia and/or requiring a platelet transfusion on 2 separate days within a 7-day period, or any grade 4 hematologic toxicity except lymphopenia. Non-hematologic DLTs included any grade 4 non-hematologic toxicity, any grade 3 non-hematologic toxicity with some exceptions (e.g., nausea and vomiting of < 5 days; diarrhea and/or electrolyte disturbances which have not been maximally treated; AST/ALT elevation that returns to levels meeting eligibility criteria within 7 days of study drug interruption and does not recur upon restarting drug), or any grade 2 non-hematologic toxicity that persists for > 7 days and is considered medically significant or sufficiently intolerable by patients requires treatment interruption.
Time Frame: 4 weeks
Population: Patients who received at least one dose of palbociclib were included in the analysis. One patient in stratum II dose level 2 who withdrew prior to beginning protocol therapy was excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2)
Number analyzed (Participants) | 3 | 12 | 6 | 4 | 9
Participants | 0 | 2 | 2 | 0 | 1

4. Primary Outcome: Single Dose Apparent Volume of Central Compartment (Vc/F)
Description: On day 1 of course 1, series blood samples for palbociclib pharmacokinetic studies were collected at pre-dose, 0.5, 1, 2, 4, 8 (±1), 10 (±0.5) optional, 24 (±4), 48 (±4) hours after the oral dose of palbociclib. Apparent volume of central compartment (Vc/F) was estimated using a non-compartmental method.
Time Frame: Up to day 3
Population: Patients with blood samples collected for pharmacokinetic studies on days 1-3 of course 1 were included.
Measure: Median (Full Range); unit: L/m^2
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2)
Number analyzed (Participants) | 3 | 12 | 6 | 4 | 9
L/m^2 | 672 [622 to 1189] | 741 [562 to 1856] | 708 [601 to 819] | 847 [373 to 1153] | 850 [398 to 3653]

5. Primary Outcome: Single Dose Elimination Rate Constant (Ke)
Description: On day 1 of course 1, series blood samples for palbociclib pharmacokinetic studies were collected at pre-dose, 0.5, 1, 2, 4, 8 (±1), 10 (±0.5) optional, 24 (±4), 48 (±4) hours after the oral dose of palbociclib. Elimination rate constant (Ke) was estimated using a non-compartmental method.
Time Frame: Up to day 3
Population: Patients with blood samples collected for pharmacokinetic studies on days 1-3 of course 1 were included.
Measure: Median (Full Range); unit: per hour
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2)
Number analyzed (Participants) | 3 | 12 | 6 | 4 | 9
per hour | 0.053 [0.045 to 0.055] | 0.053 [0.030 to 0.070] | 0.048 [0.023 to 0.083] | 0.051 [0.031 to 0.070] | 0.051 [0.014 to 0.097]

6. Primary Outcome: Single Dose Half-life (t1/2)
Description: On day 1 of course 1, series blood samples for palbociclib pharmacokinetic studies were collected at pre-dose, 0.5, 1, 2, 4, 8 (±1), 10 (±0.5) optional, 24 (±4), 48 (±4) hours after the oral dose of palbociclib. Half-life (t1/2) was estimated using a non-compartmental method.
Time Frame: Up to day 3
Population: Patients with blood samples collected for pharmacokinetic studies on days 1-3 of course 1 were included.
Measure: Median (Full Range); unit: hour
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2)
Number analyzed (Participants) | 3 | 12 | 6 | 4 | 9
hour | 13.0 [12.5 to 15.5] | 13.0 [9.9 to 22.8] | 14.6 [8.4 to 29.8] | 13.8 [10.0 to 22.0] | 13.5 [7.1 to 48.7]

7. Primary Outcome: Single Dose Apparent Oral Clearance (CL/F)
Description: On day 1 of course 1, series blood samples for palbociclib pharmacokinetic studies were collected at pre-dose, 0.5, 1, 2, 4, 8 (±1), 10 (±0.5) optional, 24 (±4), 48 (±4) hours after the oral dose of palbociclib. Apparent oral clearance (CL/F) was estimated using a non-compartmental method.
Time Frame: Up to day 3
Population: Patients with blood samples collected for pharmacokinetic studies on days 1-3 of course 1 were included.
Measure: Median (Full Range); unit: L/h/m^2
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2)
Number analyzed (Participants) | 3 | 12 | 6 | 4 | 9
L/h/m^2 | 35.8 [34.4 to 53.1] | 38.4 [29.3 to 72.0] | 33.7 [17.3 to 63.3] | 37.2 [16.9 to 64.3] | 24.4 [11.7 to 355.0]

8. Primary Outcome: Single Dose Area Under the Plasma Concentration Time Curve (AUC)
Description: On day 1 of course 1, series blood samples for palbociclib pharmacokinetic studies were collected at pre-dose, 0.5, 1, 2, 4, 8 (±1), 10 (±0.5) optional, 24 (±4), 48 (±4) hours after the oral dose of palbociclib. Area under the plasma concentration time curve (AUC) was estimated using a non-compartmental method.
Time Frame: Up to day 3
Population: Patients with blood samples collected for pharmacokinetic studies on days 1-3 of course 1 were included.
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2)
Number analyzed (Participants) | 3 | 12 | 6 | 4 | 9
h*ng/mL | 1156 [810 to 1164] | 1743 [892 to 2537] | 2407 [1485 to 3252] | 1289 [747 to 2834] | 2538 [189 to 2951]

9. Primary Outcome: Steady State Apparent Volume of Central Compartment (Vc/F)
Description: On day 21 of course 1, series blood samples for palbociclib pharmacokinetic studies were collected at pre-dose, 1, 2, 4, 8 (±1), 10 (±0.5) optional, and 24 (±4) hours after the dose. Apparent volume of central compartment (Vc/F) was estimated using a non-compartmental method.
Time Frame: Up to day 22
Population: Patients with blood samples collected for pharmacokinetic studies on days 21-22 of course 1 were included.
Measure: Median (Full Range); unit: L/m^2
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2)
Number analyzed (Participants) | 2 | 10 | 3 | 4 | 8
L/m^2 | 491 [465 to 517] | 449 [282 to 1560] | 442 [383 to 501] | 705 [250 to 1308] | 458 [247 to 919]

10. Primary Outcome: Steady State Elimination Rate Constant (Ke)
Description: On day 21 of course 1, series blood samples for palbociclib pharmacokinetic studies were collected at pre-dose, 1, 2, 4, 8 (±1), 10 (±0.5) optional, and 24 (±4) hours after the dose. Elimination rate constant (Ke) was estimated using a non-compartmental method.
Time Frame: Up to day 22
Population: Patients with blood samples collected for pharmacokinetic studies on days 21-22 of course 1 were included.
Measure: Median (Full Range); unit: per hour
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2)
Number analyzed (Participants) | 2 | 10 | 3 | 4 | 8
per hour | 0.052 [0.041 to 0.066] | 0.050 [0.017 to 0.110] | 0.062 [0.054 to 0.071] | 0.032 [0.024 to 0.049] | 0.039 [0.032 to 0.074]

11. Primary Outcome: Steady State Half-life (t1/2)
Description: On day 21 of course 1, series blood samples for palbociclib pharmacokinetic studies were collected at pre-dose, 1, 2, 4, 8 (±1), 10 (±0.5) optional, and 24 (±4) hours after the dose. Half-life (t1/2) was estimated using a non-compartmental method.
Time Frame: Up to day 22
Population: Patients with blood samples collected for pharmacokinetic studies on days 21-22 of course 1 were included.
Measure: Median (Full Range); unit: hour
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2)
Number analyzed (Participants) | 2 | 10 | 3 | 4 | 8
hour | 13.7 [10.5 to 16.9] | 13.7 [6.5 to 41.6] | 11.3 [9.8 to 12.8] | 23.1 [14.2 to 29.4] | 17.9 [9.4 to 21.4]

12. Primary Outcome: Steady State Apparent Oral Clearance (CL/F)
Description: On day 21 of course 1, series blood samples for palbociclib pharmacokinetic studies were collected at pre-dose, 1, 2, 4, 8 (±1), 10 (±0.5) optional, and 24 (±4) hours after the dose. Apparent oral clearance (CL/F) was estimated using a non-compartmental method.
Time Frame: Up to day 22
Population: Patients with blood samples collected for pharmacokinetic studies on days 21-22 of course 1 were included.
Measure: Median (Full Range); unit: L/h/m^2
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2)
Number analyzed (Participants) | 2 | 10 | 3 | 4 | 8
L/h/m^2 | 26.6 [19.0 to 34.2] | 25.8 [12.3 to 101.0] | 28.1 [20.8 to 35.3] | 17.0 [9.7 to 64.0] | 16.1 [12.1 to 62.4]

13. Primary Outcome: Steady State Area Under the Plasma Concentration Time Curve (AUC)
Description: On day 21 of course 1, series blood samples for palbociclib pharmacokinetic studies were collected at pre-dose, 1, 2, 4, 8 (±1), 10 (±0.5) optional, and 24 (±4) hours after the dose. Area under the plasma concentration time curve (AUC) was estimated using a non-compartmental method.
Time Frame: Up to day 22
Population: Patients with blood samples collected for pharmacokinetic studies on days 21-22 of course 1 were included.
Measure: Median (Full Range); unit: h*ng/mL
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2)
Number analyzed (Participants) | 2 | 10 | 3 | 4 | 8
h*ng/mL | 1211 [972 to 1450] | 2143 [521 to 4070] | 2193 [1520 to 3168] | 1410 [559 to 3301] | 2359 [952 to 4253]

14. Secondary Outcome: Number of Subjects With Objective Responses
Description: Objective responses included complete response (CR) and partial response (PR).
Time Frame: Up to 2 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2)
Number analyzed (Participants) | 3 | 12 | 6 | 4 | 9
Participants | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Association Between Neutropenia and Single Dose Palbociclib AUC
Description: Neutrophil count decreased adverse events observed in course 1 that were at least possibly attributable to palbociclib were included in analysis. Based on the highest toxicity grade reported, all participants, irrespective of their dose level or stratum, were combined and classified into three categories: 0 = no toxicity reported, 1 = grade 1 or 2, and 2 = grade 3 or 4. Association between neutrophil count decreased and single dose palbociclib AUC for all participants was examined.
Time Frame: Up to approximately 4 weeks
Population: It was pre-specified that data from all participants from different dose levels and strata were combined to calculate an association between neutropenia and single dose AUC for all participants. Of 35 patients enrolled, one patient in stratum II withdrew prior to protocol therapy and was excluded.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- All Patients: All 34 patients who had course 1 single dose palbociclib AUC data available were included in analysis. Patients were classified into no neutropenia (n = 9), grade 1 or 2 neutropenia (n = 7), and grade 3 or 4 neutropenia (n = 18).
Arm/Group | All Patients
Number analyzed (Participants) | 34
h*ng/mL
  No neutropenia: number analyzed (Participants) | 9
  No neutropenia | 1424.4 (966.3)
  Grade 1 or 2 neutropenia: number analyzed (Participants) | 7
  Grade 1 or 2 neutropenia | 2166.3 (797.8)
  Grade 3 or 4 neutropenia: number analyzed (Participants) | 18
  Grade 3 or 4 neutropenia | 1937.6 (621.8)
Statistical Analysis 1: Comparison: All Patients; Test type: Other — Ordinal logistic regression model was built for outcome neutropenia (0/1/2). Explanatory variable AUC was transformed by dividing by 100; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.97 to 1.15]

16. Secondary Outcome: Association Between Lymphopenia and Single Dose Palbociclib AUC
Description: Lymphocyte count decreased adverse events observed in course 1 that were at least possibly attributable to palbociclib were included in analysis. Based on the highest toxicity grade reported, all participants, irrespective of their dose level or stratum, were combined and classified into three categories: 0 = no toxicity reported, 1 = grade 1 or 2, and 2 = grade 3 or 4. Association between Lymphocyte count decreased and single dose palbociclib AUC for all participants was examined.
Time Frame: Up to approximately 4 weeks
Population: It was pre-specified that data from all participants from different dose levels and strata were combined to calculate an association between lymphopenia and single dose AUC for all participants. Of 35 patients enrolled, one patient in stratum II withdrew prior to protocol therapy and was excluded.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- All Patients: All 34 patients who had course 1 single dose palbociclib AUC data available were included in analysis. Patients were classified into no lymphopenia (n = 17), grade 1 or 2 lymphopenia (n = 10), and grade 3 or 4 lymphopenia (n = 7).
Arm/Group | All Patients
Number analyzed (Participants) | 34
h*ng/mL
  No lymphopenia: number analyzed (Participants) | 17
  No lymphopenia | 1727.5 (882.6)
  Grade 1 or 2 lymphopenia: number analyzed (Participants) | 10
  Grade 1 or 2 lymphopenia | 1837.9 (592.7)
  Grade 3 or 4 lymphopenia: number analyzed (Participants) | 7
  Grade 3 or 4 lymphopenia | 2159.0 (793.7)
Statistical Analysis 1: Comparison: All Patients; Test type: Other — Ordinal logistic regression model was built for outcome lymphopenia (0/1/2). Explanatory variable AUC was transformed by dividing by 100; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.97 to 1.15]

17. Secondary Outcome: Association Between Leukopenia and Single Dose Palbociclib AUC
Description: White blood cell count decreased adverse events observed in course 1 that were at least possibly attributable to palbociclib were included in analysis. Based on the highest toxicity grade reported, all participants, irrespective of their dose level or stratum, were combined and classified into three categories: 0 = no toxicity reported, 1 = grade 1 or 2, and 2 = grade 3 or 4. Association between white blood cell count decreased and single dose palbociclib AUC for all participants was examined.
Time Frame: Up to approximately 4 weeks
Population: It was pre-specified that data from all participants from different dose levels and strata were combined to calculate an association between leukopenia and single dose AUC for all participants. Of 35 patients enrolled, one patient in stratum II withdrew prior to protocol therapy and was excluded.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- All Patients: All 34 patients who had course 1 single dose palbociclib AUC data available were included in analysis. Patients were classified into no leukopenia (n = 8), grade 1 or 2 leukopenia (n = 17), and grade 3 or 4 leukopenia (n = 9).
Arm/Group | All Patients
Number analyzed (Participants) | 34
h*ng/mL
  No leukopenia: number analyzed (Participants) | 8
  No leukopenia | 1420.3 (955.1)
  Grade 1 or 2 leukopenia: number analyzed (Participants) | 17
  Grade 1 or 2 leukopenia | 1879.6 (682.6)
  Grade 3 or 4 leukopenia: number analyzed (Participants) | 9
  Grade 3 or 4 leukopenia | 2171.6 (712.9)
Statistical Analysis 1: Comparison: All Patients; Test type: Other — Ordinal logistic regression model was built for outcome leukopenia (0/1/2). Explanatory variable AUC was transformed by dividing by 100; Odds Ratio (OR) = 1.10, 95% CI 2-sided [1.01 to 1.20]

18. Other Pre Specified Outcome: Number of Subjects With Cyclin-dependent Kinase-4 (CDK4) Copy Number Variations
Description: CDK4 is a key component in signaling pathways inside normal cells and cancer cells. CDK4 copy number variations were to be assessed by array comparative genomic hybridization in available tumor tissues from consenting patients.
Time Frame: At enrollment
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Number of Subjects With Cyclin-dependent Kinase-6 (CDK6) Copy Number Variations
Description: CDK6 is a key component in signaling pathways inside normal cells and cancer cells. CDK6 copy number variations were to be assessed by array comparative genomic hybridization in available tumor tissues from consenting patients.
Time Frame: At enrollment
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Number of Subjects With Cyclin D1 Copy Number Variations
Description: Cyclin D1 is a key component in signaling pathways inside normal cells and cancer cells. Cyclin D1 copy number variations were to be assessed by array comparative genomic hybridization in available tumor tissues from consenting patients.
Time Frame: At enrollment
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Number of Subjects With Cyclin D2 Copy Number Variations
Description: Cyclin D2 is a key component in signaling pathways inside normal cells and cancer cells. Cyclin D2 copy number variations were to be assessed by array comparative genomic hybridization in available tumor tissues from consenting patients.
Time Frame: At enrollment
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Number of Subjects With Cyclin D3 Copy Number Variations
Description: Cyclin D3 is a key component in signaling pathways inside normal cells and cancer cells. Cyclin D3 copy number variations were to be assessed by array comparative genomic hybridization in available tumor tissues from consenting patients.
Time Frame: At enrollment
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Number of Subjects With Ink4a-ARF Loss Copy Number Variations
Description: Ink4a-ARF is a key component in signaling pathways inside normal cells and cancer cells. Ink4a-ARF loss copy number variations were to be assessed by array comparative genomic hybridization in available tumor tissues from consenting patients.
Time Frame: At enrollment
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Polymorphisms in Efflux-transporter Proteins P-glycoprotein (P-gp; ABCB1)
Description: Polymorphisms in ABCB1 encode for efflux-transporter proteins P-glycoprotein (P-gp), for which palbociclib has been shown as a substrate. Genomic DNA was to be isolated from peripheral blood samples from consenting patients to determine ABCB1 polymorphisms.
Time Frame: At enrollment
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Polymorphisms in Breast Cancer Resistance Protein (BCRP; ABCG2)
Description: Polymorphisms in ABCG2 encode for BCRP, for which palbociclib has been shown as a substrate. Genomic DNA was to be isolated from peripheral blood samples from consenting patients to determine ABCG2 polymorphisms.
Time Frame: At enrollment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 2 years after starting treatment
Description: Adverse events (AEs) were graded using CTCAE v4.0. AEs collected per protocol included: a) grade 1 and 2 AEs if attribution was at least possibly related to palbociclib and b) all grade 3+ AEs on treatment and within 30 days off treatment. AEs that were at least possibly attributable to palbociclib were summarized in SAE and Other AE tables below. All mortality on this study were due to disease. One patient in stratum II dose level 2 withdrew prior to protocol therapy and was not at risk.
Arm/Group | Stratum I, Dose Level 1 (50 mg/m2) | Stratum I, Dose Level 2 (75 mg/m2) | Stratum I, Dose Level 3 (95 mg/m2) | Stratum II, Dose Level 1 (50 mg/m2) | Stratum II, Dose Level 2 (75mg/m2)
All-Cause Mortality (participants affected / at risk) | 0/3 | 3/12 | 1/6 | 1/4 | 1/9
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/12 | 1/6 | 0/4 | 0/9
Other Adverse Events (participants affected / at risk) | 3/3 | 12/12 | 5/6 | 4/4 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum I, Dose Level 1 (50 mg/m2) (N=3) | Stratum I, Dose Level 2 (75 mg/m2) (N=12) | Stratum I, Dose Level 3 (95 mg/m2) (N=6) | Stratum II, Dose Level 1 (50 mg/m2) (N=4) | Stratum II, Dose Level 2 (75mg/m2) (N=9)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum I, Dose Level 1 (50 mg/m2) (N=3) | Stratum I, Dose Level 2 (75 mg/m2) (N=12) | Stratum I, Dose Level 3 (95 mg/m2) (N=6) | Stratum II, Dose Level 1 (50 mg/m2) (N=4) | Stratum II, Dose Level 2 (75mg/m2) (N=9)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 5 (6) | 2 (3) | 4 (8) | 6 (11)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - other, specify (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (6) | 1 (1) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - other, specify (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 3 (10) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (4) | 0 (0) | 1 (1) | 2 (4)
Fatigue (General disorders) | 1 (1) | 5 (5) | 1 (1) | 1 (1) | 3 (3)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (3)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Investigations - other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (3) | 8 (44) | 3 (3) | 2 (10) | 4 (8)
Neutrophil count decreased (Investigations) | 1 (3) | 10 (54) | 3 (6) | 4 (13) | 7 (25)
Platelet count decreased (Investigations) | 1 (1) | 6 (23) | 3 (4) | 2 (10) | 5 (13)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 2 (3) | 10 (57) | 5 (10) | 4 (15) | 7 (22)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Informed Consent Form (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/61/NCT02255461/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/61/NCT02255461/Prot_SAP_002.pdf